CLINICAL TRIAL: NCT01460030
Title: An Intra-individual Titration Study of KRN1493 for the Treatment of Hypercalcemia in Patients With Parathyroid Carcinoma or Intractable Primary Hyperparathyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: KRN1493-101
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Parathyroid Carcinoma; Hypercalcemia; Primary Hyperparathyroidism
Keywords: Hypercalcemia in patients with parathyroid carcinoma or intractable PHPT
MeSH Terms: conditions — Parathyroid Neoplasms; Hypercalcemia; Hyperparathyroidism, Primary | interventions — Cinacalcet

ARMS (1):
- KRN1493 (Experimental)
  Interventions: Drug: Cinacalcet HCl

INTERVENTIONS:
Drug: Cinacalcet HCl — Oral administration

SUMMARY:
This is an intra-individual titration study of KRN1493 to evaluate the safety and efficacy of KRN1493 for the treatment of hypercalcemia in patients with parathyroid carcinoma or intractable primary hyperparathyroidism (PHPT).

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet any one of the following. Patients with a diagnosis of parathyroid carcinoma and corrected serum calcium > 11.3 mg/dL at the latest screening test. Patients with intractable PHPT (defined as follows: impossible to localize parathyroid tumor before initial surgery or in relapse after surgery, or impossible to perform parathyroidectomy (PTx) for complications, and corrected serum calcium is > 12.5 mg/dL at the screening test).
* Patients who provided their voluntary written informed consent to participate in the study.

Exclusion Criteria:

* Patients diagnosed with malignant tumor except for parathyroid carcinoma, nonmelanoma skin cancer, and carcinoma in situ of the cervix within 5 years before enrollment.
* Patients receiving anticancer chemotherapy except for the treatment of parathyroid carcinoma.
* Patients diagnosed with hypercalcemia associated with malignant tumors other than parathyroid carcinoma.
* Patients who had hypersensitivities to cinacalcet HCl preparations or vehicles.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Corrected serum calcium

SECONDARY OUTCOMES:
Serum intact parathyroid hormone

CONTACTS AND LOCATIONS:
Locations (1):
- Sendai, Japan